CLINICAL TRIAL: NCT01563679
Title: Prospective Analysis of Percutaneous Ablations for Cancer Treatment
Brief Title: Analysis of Percutaneous Ablations for Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hyun Kevin Kim, Director of Interventional Radiology and Image-guided Medicine, Emory University
Other Study IDs: IRB00054905; RAD2160-11 (Other: Other)
Record Dates: First submitted 2012-03-12; First posted 2012-03-27 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Cancer
Keywords: cancer; locoregional therapies; RFA; Cryoablation; Microwave ablation; chemical ablation; Irreversible electroporation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a study involving patients with cancer who are referred by their treating physician for percutaneous locoregional therapies.

Patient's clinical and radiology findings, pathology findings, survival, treatment responses, and complications after their locoregional therapy will be studied.

DETAILED DESCRIPTION:
The efficacy of the percutaneous and transarterial treatments for solid tumors will be studied. Prospective study on patients who receive percutaneous locoregional therapies, including radiofrequency ablation (RFA), cryoablation, microwave ablation, IRE and chemical ablation for treatment of cancer will be performed.

Preoperative clinic chart, procedure note, postoperative chart, pre- and post-operative CT, MRI or Ultrasound, angiographic findings, biopsy results and pathologic findings, will be reviewed. Patient survival, treatment responses, complications after the therapy will be collected from clinic visits and clinical encounters.

Patient overall performance status before and after procedures will be assessed using the Quality of Life questionnaire (SF-36™ Health Survey).

ELIGIBILITY:
Inclusion Criteria:

* 18yrs of age
* Cancer diagnosis
* Candidate for Locoregional therapy
* Willingness to sign informed consent

Exclusion Criteria:

* Unable to sign informed consent
* Patients not eligible for locoregional therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo ablative therapy procedures, in the Interventional Radiology department as part of a clinical treatment for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Effect of percutaneous and transarterial treatments for cancer in quality of life | 1 year
  Patients will complete the QOL questionnare during their follow up visits after procedure. 1 month, 3 months, 6 months and 1 year.

SECONDARY OUTCOMES:
response rate to percutaneous and transarterial treatment for cancer | 1 month, 3 months, 6 months, 1 year.
  Patients will be followed up 1, 3, 6 and 1year intervals after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun S Kim, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Altanta, Georgia, United States